CLINICAL TRIAL: NCT04425005
Title: Effect of Home-based Exercise Training Program During the Covid-19 Pandemic in Post-bariatric Patients: A Randomized Controlled Trial
Brief Title: Home-based Exercise Training During Covid-19 Pandemic in Post-bariatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21056813.3.0000.0068
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Bariatric Surgery; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention)
- Exercise training group (Experimental)
  Interventions: Other: Home-based exercise

INTERVENTIONS:
Other: Home-based exercise — Home-based exercise training, supervised by videoconference.
  Arms: Exercise training group

SUMMARY:
The aim of this study is to assess the effect of a home-based exercise training during social isolation due to covid-19 pandemic in patients who undertook bariatric surgery.

DETAILED DESCRIPTION:
Eligible patients will be invited to participate in the study by phone call. The research team will visit the included patients. All patients giving the written consent will perform the following tests before being randomly allocated into exercise training or control: 1) blood pressure; 2) anthropometric measures; 3) blood sampling; 4) handgrip test; 5) sit and stand test; 6) exercise capacity; 7) nutritional recalls and 8) health-related questionnaires. Patients will be randomized in a 1:1 ratio to control group (will receive information to keep active and eating healthy) or exercise training group (will receive a telemonitored exercise program through video conference, three times a week, during 3 months). Following 3 months of intervention, the outocomes will be re-assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women submitted to bariatric surgery in the last 12 months.
* Not engaged in regular exercise training programs.

Exclusion Criteria:

* Patients with >12 months of post-operatory period.
* Patients with diagnosed mental disorders.
* Patients with physical limitations or not allowed by the physician to exercise.
* Patients infected with Covid-19 at the time of data collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline on waist circumference at 3 months of follow-up. | Baseline and 3 months
  Waist circumference will be measured using a steel measuring tape to the nearest 0.1cm at the high point of the iliac crest at minimal respiration.

SECONDARY OUTCOMES:
Change from baseline on cardiometabolic risk factor at 3 months of follow-up. | Baseline and 3 months
  Cardiometabolic risk will be calculated using mean blood pressure, fasting triglycerides, HDL, waist circumference and fasting glucose. These outocomes will be presented separately as well.
Change from baseline on cardiopulmonary fitness at 3 months of follow-up. | Baseline and 3 months
  Cardiopulmonary fitness will be assessed by a validated two-minutes step test.
Change from baseline on quality of life at 3 months of follow up. | Baseline and 3 months
  Will be evaluated by the SF-36 health survey questionnaire.
Change from baseline on Physical activity levels at 3 months of follow up. | Baseline and 3 months follow-up.
  Will be evaluated by the International Physical Activity Questionnaire.
Change from baseline on dietary intake at 3 months of follow up. | Baseline and 3 months
  Will be assessed by 24 hours food intake recall.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, Principal Investigator — HC FMUSP
Locations (1):
- Univsersity of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No